CLINICAL TRIAL: NCT04000763
Title: Superficial Peroneal Nerve Neuromodulation for Non-Obstructive Urinary Retention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christopher J Chermansky, MD (Other)
Collaborators: Society of Urodynamics, Female Pelvic Medicine & Urogenital Reconstruction (Other); University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor-Investigator, Christopher J Chermansky, MD, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY19010062
Record Dates: First submitted 2019-05-23; First posted 2019-06-27 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Urinary Retention; Urinary Bladder, Underactive
Keywords: Bladder
MeSH Terms: conditions — Urinary Retention; Urinary Bladder, Underactive

STUDY DESIGN:
Intervention Model Description: All experiments proposed in this grant application will be performed in female non-obstructive urinary retention patients. We chose not to study male patients in this study given the need to exclude bladder outlet obstruction from benign prostatic hyperplasia (BPH), an evaluation that is invasive and costly.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Transcutaneous Nerve Stimulator(TENS) (Experimental): Adult females who have difficulty emptying their bladder due to non-obstructive urinary retention or because of an under-active bladder will be given transcutaneous nerve stimulation (TENS) therapy.
  Interventions: Device: superficial peroneal nerve stimulation

INTERVENTIONS:
Device: superficial peroneal nerve stimulation — A commercially available FDA-approved transcutaneous electrical nerve stimulator (TENS) and skin surface electrodes will be used to stimulate the foot. The electrodes will be attached to the dorsal surface of the foot and a sock will be placed over the foot to prevent detachment of the electrodes. Based on our animal studies, foot stimulation parameters of 2 Hz frequency and 0.2 ms pulse width will be used at the maximal intensity comfortable for each patient. It is expected that superficial peroneal nerve stimulation in patients can increase bladder sensation so that micturition can be initiated at a small bladder volume, or it can initiate bladder contraction at a small bladder volume and enhance the contraction or prolong the duration of contraction. Any of these excitatory effects, if occurs in human patients, will certainly improve the condition of non-obstructive urinary retention.

SUMMARY:
Millions of Americans are suffering from underactive bladder (UAB). The impact of severe UAB, i.e. non-obstructive urinary retention (NOUR) on quality of life is significant because current treatment for non-obstructive urinary retention requires intermittent self-catheterization or an indwelling suprapubic catheter. Currently an effective drug for non-obstructive urinary retention does not exist. It is a therapeutic challenge for clinicians to successfully treat non-obstructive urinary retention. Sacral neuromodulation has been approved by the FDA since 1999 to treat non-obstructive urinary retention. It achieves >50% improvement in bladder emptying (reducing the frequency of self-catheterization or increasing voided volume) in just over half of the patients. Sacral neuromodulation requires surgical implantation of a stimulator and a lead with 4 electrodes. The surgery and implant are invasive and expensive, preventing a broad application of this effective therapy to many non-obstructive urinary retention patients. The goal of this study is to develop a novel non-invasive neuromodulation therapy for non-obstructive urinary retention as an alternative. Specifically, the investigators will explore the possibility to translate into humans a recent discovery in cats of an excitatory reflex from the superficial peroneal nerve to the bladder to treat non-obstructive urinary retention. Therefore, in this study the investigators propose to develop a non-invasive, transcutaneous neuromodulation therapy for non-obstructive urinary retention that can be administered at home.

DETAILED DESCRIPTION:
Hypothesis: Electrical stimulation of the superficial peroneal nerve using transcutaneous skin electrodes attached on the dorsal foot can treat non-obstructive urinary retention either by enhancing bladder sensation thereby reducing bladder volume needed for initiating voiding and/or by enhancing bladder contraction, thereby increasing voiding efficiency and reducing post-void residual (PVR) volume.

Rationale: The investigators conducted preliminary studies in cats that have demonstrated an excitatory reflex to the bladder elicited by stimulation of afferent axons in the superficial peroneal nerve. Activating this excitatory reflex in cats reduced bladder capacity (the minimal volume for initiating a micturition reflex), enhanced bladder contractions and overcame bladder inhibition emanating from somatic (tibial) afferent activation. Since the superficial peroneal nerve innervates the dorsal skin of the foot in humans, it can be stimulated non-invasively by skin surface electrodes. Transcutaneous stimulation of this nerve, should it prove efficacious, would likely be more acceptable to patients with non-obstructive urinary retention (NOUR) than invasive sacral neuromodulation therapy. Therefore, in this study, the investigators propose to test the superficial peroneal nerve neuromodulation in non-obstructive urinary retention patients.

Specific Aim: Determine the efficacy of superficial peroneal nerve stimulation (SPNS) in the treatment of patients with non-obstructive urinary retention using skin electrodes attached to the dorsal surface of the foot.

Rationale: Based on a preliminary discovery in cats, the investigators propose to further investigate the effect of superficial peroneal nerve stimulation (SPNS) on voiding efficiency, post-void residual (PVR) volume, and bladder capacity (voided volume + post-void residual) in patients with non-obstructive urinary retention. A reduced bladder capacity indicates more normal bladder filling sensations, thereby allowing voiding at more normal volumes. The investigators plan to test superficial peroneal nerve stimulation in 10 non-obstructive urinary retention patients by collecting voiding diary during a 3-week period. Baseline voiding diary will be collected during the first week before superficial peroneal nerve stimulation initiation. During the second week, superficial peroneal nerve stimulation will be administered to each patient for 3 hours/day before sleep and it will also be administered immediately prior and throughout each void. The 3-hour stimulation is designed to modulate bladder sensory pathways to enhance bladder sensation, thereby reducing the bladder volume required to initiate voiding. The acute stimulation during each void is designed to enhance bladder contraction, thereby increasing voiding efficiency and reducing post-void residual. During the third week, superficial peroneal nerve stimulation will not be applied, and a voiding diary will be collected to determine any post-stimulation effect. Since the superficial peroneal nerve is a cutaneous nerve innervating the skin of the dorsal foot, superficial peroneal nerve stimulation will be applied non-invasively by attaching skin surface electrodes to the dorsal side of the foot.

ELIGIBILITY:
Inclusion Criteria:

Able to provide informed consent

1. 18 years of age and older
2. Clinically diagnoses as non-obstructive urinary retention
3. Post Void Residual of 300 mL or greater
4. Currently using daily self-catheterization to empty the bladder
5. Capable of using the toilet independently without difficulty
6. Capable and willing to follow all study-related procedures

Exclusion Criteria:

1. Neurologic diagnosis (including diabetes mellitus)
2. Surgery within one year of screening for urinary outlet obstruction
3. Pregnant or planning to become pregnant during study duration
4. OnabotulinumtoxiA use in bladder or pelvic floor muscles with the past year
5. Pacemaker or implantable defibrillator
6. Current Urinary tract or vaginal infections
7. Current Interstim use
8. Current Percutaneous tibial nerve stimulation (PTNS) or transcutaneous electrical nerve stimulation (TENS) use in pelvis or back or legs
9. Investigational drug/ device therapy with the past 4 weeks,
10. Participation in any clinical investigation involving or impacting gynecologic or urinary function with the past 4 weeks,
11. Previous surgery of or damage to the foot or nerves in the foot and leg.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Number of voids per subject in 24 hours. | 3 weeks
  Counted using a patient voiding diary both before and after superficial peroneal nerve stimulation.
Number of catheterizations per subject in 24 hours. | 3 weeks
  Counted using a patient voiding diary both before and after superficial peroneal nerve stimulation.
Volume of urine per void. | 3 weeks
  Calculated in millimeters both before and after peroneal nerve stimulation.
Catheterized Post Void Residual volume | 3 weeks
  Calculated in millimeters both before and after peroneal nerve stimulation.
Bladder Voiding efficiency | 3 weeks
  Pre voiding and post voiding ratio that reflects bladder contractility
Bladder capacity | 3 weeks
  Calculated by adding the voided volume to the post residual catheterization volume, in milliliters

SECONDARY OUTCOMES:
Efficacy of Foot Stimulation | 2 weeks
  Difference in millimeters of bladder emptying capacity from week 2 to baseline
Efficacy of Foot Stimulation | 3 weeks
  Difference in millimeters of bladder emptying capacity from week 3 to baseline
Post-stimulation effect | 1 week
  Difference in millimeters of bladder emptying capacity from week 2 to week 3.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Chermansky, MD, Study Director — University of Pittsburgh
Locations (1):
- UPMC Urology, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data and methods will be shared with other investigators upon signed data use agreements and assurance of Institutional Review Board approval.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After all data is collected and analyzed.
Access Criteria: Data Use Agreement Institutional Review Board approval.

REFERENCES:
- [Background] 26872574
- [Background] Juszczak K, Drewa T. Pharmacotherapy in detrusor underactivity: A new challenge for urologists and pharmacologists (from lab to clinic). Pharmacol Rep. 2016 Aug;68(4):703-6. doi: 10.1016/j.pharep.2016.03.007. Epub 2016 Mar 19. PMID 27110877
- [Background] Kessler TM, Fowler CJ. Sacral neuromodulation for urinary retention. Nat Clin Pract Urol. 2008 Dec;5(12):657-66. doi: 10.1038/ncpuro1251. Epub 2008 Nov 11. PMID 19002127
- [Background] De Ridder D, Ost D, Bruyninckx F. The presence of Fowler's syndrome predicts successful long-term outcome of sacral nerve stimulation in women with urinary retention. Eur Urol. 2007 Jan;51(1):229-33; discussion 233-4. doi: 10.1016/j.eururo.2006.06.031. Epub 2006 Jul 10. PMID 16860462
- [Background] Faraj K, Doo F, Boura J, Vereecke A, Chancellor MB. A cross-sectional study in the USA of the epidemiology and quality of life of underactive bladder symptoms. Int Urol Nephrol. 2016 Nov;48(11):1797-1802. doi: 10.1007/s11255-016-1382-0. Epub 2016 Jul 29. PMID 27473156
- [Background] Abarbanel J, Marcus EL. Impaired detrusor contractility in community-dwelling elderly presenting with lower urinary tract symptoms. Urology. 2007 Mar;69(3):436-40. doi: 10.1016/j.urology.2006.11.019. PMID 17382138
- [Background] Goodwin RJ, Swinn MJ, Fowler CJ. The neurophysiology of urinary retention in young women and its treatment by neuromodulation. World J Urol. 1998;16(5):305-7. doi: 10.1007/s003450050072. PMID 9833308
- [Background] Jonas U, Fowler CJ, Chancellor MB, Elhilali MM, Fall M, Gajewski JB, Grunewald V, Hassouna MM, Hombergh U, Janknegt R, van Kerrebroeck PE, Lylcklama a Nijeholt AA, Siegel SW, Schmidt RA. Efficacy of sacral nerve stimulation for urinary retention: results 18 months after implantation. J Urol. 2001 Jan;165(1):15-9. doi: 10.1097/00005392-200101000-00004. PMID 11125353
- [Background] Yu M, Uy J, Jiang X, Li X, Jones C, Shen B, Wang J, Roppolo JR, de Groat WC, Tai C. An excitatory reflex from the superficial peroneal nerve to the bladder in cats. Am J Physiol Renal Physiol. 2017 Nov 1;313(5):F1161-F1168. doi: 10.1152/ajprenal.00265.2017. Epub 2017 Aug 30. PMID 28855188
- [Background] Tai C, Shen B, Chen M, Wang J, Roppolo JR, de Groat WC. Prolonged poststimulation inhibition of bladder activity induced by tibial nerve stimulation in cats. Am J Physiol Renal Physiol. 2011 Feb;300(2):F385-92. doi: 10.1152/ajprenal.00526.2010. Epub 2010 Nov 24. PMID 21106856